CLINICAL TRIAL: NCT00212823
Title: AXERT® 12.5mg Time vs Intensity Migraine Study (AIMS): An Open-label Multicenter Trial to Evaluate the Efficacy of Almotriptan Malate (AXERT®) 12.5 Milligram Intervention at Onset of Migraine Pain
Brief Title: The Effectiveness of Almotriptan Malate (AXERT®) 12.5 Milligrams When Taken at the Onset of Migraine Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004708
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — almotriptan

INTERVENTIONS:
Drug: almotriptan malate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of AXERT when treating a migraine at the onset of headache pain, as compared to treating a migraine only after the headache pain has reached at least moderate intensity..

DETAILED DESCRIPTION:
AXERT has been approved by the FDA for the treatment of migraine headache with or without aura in adults. Early treatment of a migraine headache, independent of headache pain intensity symptoms, may provide the optimal therapeutic response. This is a multi-center, open label study to test the efficacy (effectiveness) and tolerability of AXERT when treating a migraine at the onset of headache pain versus treating a migraine only after the headache pain has reached at least moderate intensity. Patients will self-administer 12.5 milligrams of AXERT for the treatment of 2 migraine headaches. Centers will be randomly assigned to 1 of 2 treatment interventions in which patients will sequentially treat both migraine headaches with 12.5 milligrams of AXERT using either the early treatment regimen (ET; ie, at the onset of pain) or conditional treatment regimen (CT; ie, after the headache has reached at least moderate intensity). Data will be collected regarding treatment response during and after each migraine headache. For each headache, patients will record study information and data during 3 telephone calls using Interactive Voice Response System (IVRS) technology. It is expected that patients who take 12.5 milligrams of AXERT at the first sign of pain of any intensity due to a migraine headache will experience an overall shorter duration of their migraine than patients who take AXERT 12.5 mg when their migraine pain has reached at least moderate pain intensity. In addition, it is expected that almotriptan malate (AXERT®) is generally well-tolerated.

AXERT 12.5 milligram tablet orally either at the onset of migraine pain (within 1 hour of the start of a migraine-ET regimen) or when migraine pain reaches at least moderate intensity (CT regimen).

ELIGIBILITY:
Inclusion Criteria:

* History of a confirmed diagnosis of migraine headache with or without aura that meets the International Headache Society (IHS) criteria of migraine headache for at least 1 year
* Average frequency of 1 - 6 migraine headaches per month over the past 3 months
* History of migraine headaches of at least moderate pain intensity within the past year
* If taking a medication for migraine prophylaxis, taking a maintenance dose for at least 4 weeks prior to Visit 1, and remaining on a stable dose for the duration of the study
* In generally good health
* Capable of taking oral medication, perform study procedures and follow directions regarding collection of study information, e.g., subjects must be able and willing to read and comprehend written instructions, use a stopwatch, and comprehend and complete the telephone requirements, and must be willing to return to the office for a final study visit
* If female of childbearing potential, using birth control

Exclusion Criteria:

* Onset of migraine after age 50
* Chronic migraine or chronic tension-type headache defined by having 15 or more headache days per month in the previous 6 months
* Exclusively migraine aura without headache, or headaches that occur predominantly upon awakening in the morning
* Patients in whom triptans are contraindicated or who have previously discontinued AXERT therapy due to adverse events, history of substance abuse, or chronic alcohol abuse within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Actual)
Dates: Start 2004-06; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Duration of migraine pain measured from onset of pain to no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho McNeil Neurologics, Inc. Clinical Trial, Study Director — Ortho-McNeil Neurologics, Inc.

REFERENCES:
- [Result] Freitag FG, Finlayson G, Rapoport AM, Elkind AH, Diamond ML, Unger JR, Fisher AC, Armstrong RB, Hulihan JF, Greenberg SJ; AIMS Investigators. Effect of pain intensity and time to administration on responsiveness to almotriptan: results from AXERT 12.5 mg Time Versus Intensity Migraine Study (AIMS). Headache. 2007 Apr;47(4):519-30. doi: 10.1111/j.1526-4610.2007.00756.x. PMID 17445101
- See also: AXERT 12.5mg Time vs Intensity - Migraine Study (AIMS) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=919&filename=CR004708_CSR.pdf